CLINICAL TRIAL: NCT00693225
Title: Impact of Timing on the Efficacy of Omeprazole/Sodium Bicarbonate Zegerid 40 mg in Healing Reflux Esophagitis
Brief Title: Impact of Timing on the Efficacy of Zegerid 40 mg in Healing Reflux Esophagitis: A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yvonne Romero (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Yvonne Romero, Yvonne Romero, MD, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-008503
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Results first posted 2012-09-20 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-08

CONDITIONS: Erosive Esophagitis
Keywords: Erosive Esophagitis; Reflux Esophagitis; Gastroesophageal reflux disease; GERD; proton pump inhibitor; omeprazole/sodium bicarbonate
MeSH Terms: conditions — Esophagitis, Peptic; Gastroesophageal Reflux | interventions — omeprazole, sodium bicarbonate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omeprazole/sodium bicarbonate AM dose (Active Comparator): 8 weeks of therapy with omeprazole/sodium bicarbonate oral suspension 40 mg, once per day, taken in the morning
  Interventions: Drug: Omeprazole/sodium bicarbonate
- Omeprazole/sodium bicarbonate PM dose (Experimental): 8 weeks of therapy with omeprazole/sodium bicarbonate oral suspension 40 mg, once per day, taken at bedtime
  Interventions: Drug: Omeprazole/sodium bicarbonate

INTERVENTIONS:
Drug: Omeprazole/sodium bicarbonate — Omeprazole/sodium bicarbonate powder for oral suspension 40 mg was supplied in individual packets that were emptied into a small cup containing 15-30 ml (1-2 tablespoons) of water, one per day, for 8 weeks.
  Other Names: Zegerid

SUMMARY:
The purpose of this study was to determine the effect of morning versus bedtime administration of omeprazole/sodium bicarbonate (Zegerid) on endoscopic healing for patients with moderate or severe reflux esophagitis. Our hypothesis was that bedtime administration of Zegerid would be superior in healing esophagitis compared to morning administration prior to a meal.

DETAILED DESCRIPTION:
Hypothesis: The timing of administration of omeprazole/sodium bicarbonate (Zegerid) will impact nocturnal esophageal acid exposure and healing of esophagitis. Specifically, we hypothesize that omeprazole/sodium bicarbonate, taken at bedtime, will be superior in healing esophagitis compared to omeprazole/sodium bicarbonate taken in the morning.

Specific Aim: Compare the percent of subjects with moderate/severe esophagitis who achieve complete endoscopic resolution after 8 weeks of treatment (morning vs. bedtime).

Intervention: All subjects received a one-on-one educational session describing the normal physiology of the upper gastrointestinal tract, the pathophysiology of hiatal hernia and reflux esophagitis, and food stuffs that contribute to reflux, prior to their invitation to participate in the trial. Outpatients who underwent a clinically indicated esophagogastroduodenoscopy (EGD) as advised by their primary health care provider in an open-access endoscopy unit who were diagnosed with Los Angeles grade C or D erosive reflux esophagitis were invited to participate.

Omeprazole/sodium bicarbonate powder for oral suspension 40 mg was supplied in individual packets that are emptied into a small cup containing 15-30 ml (1-2 tablespoons) of water, one per day, for 8 weeks. They were asked to stir well and drink immediately then refill the cup with water and drink. Subjects assigned to morning dosing were instructed to take the medication on an empty stomach, immediately upon rising, 20 to 60 minutes prior to chewing a solid. Subjects assigned to bedtime dosing were instructed to keep the medication by their bedside; taking the medication in a standing or seated upright position immediately before turning off the lights with the intention to sleep. The subject was instructed to not use other liquids or foods for 20 minutes after taking their study medication for those allocated to morning dosing, and until the next morning for those allocated to bedtime dosing.

Gelusil™ was distributed for use as an "on demand" rescue antacid; the frequency of use was recorded with the plan to use Gelusil™ consumption as a potential confounder of omeprazole/sodium bicarbonate efficacy. Other antacids, including sodium bicarbonate, magnesium hydroxide, calcium carbonate, and sucralfate were prohibited. Subjects taking non-omeprazole proton pump inhibitors (PPIs) and/or Histamine Receptor Antagonist (HRAs) were advised to discontinue these medications while they participated in this study. No other medication was altered for this study.

After 8 weeks, a follow-up EGD was performed to assess mucosal integrity by an endoscopist blinded to the study and subject allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have either moderate to severe erosive esophagitis (Los Angeles grade C or D)
2. Subjects with esophagitis despite use of a non-omeprazole Proton Pump Inhibitor (PPI)(s) or histamine receptor antagonist (HRA) were invited to participate without a wash-out period.
3. Subjects able to return to Mayo Clinic Rochester for follow up endoscopy 8 weeks after start of study.
4. Female subjects are eligible if they are not pregnant or lactating and one of the following criteria is met:

   1. Surgically sterile (by means of hysterectomy or bilateral tubal ligation).
   2. At least one year postmenopausal (no menses for greater than or equal to 12 months).
   3. Subject is using a highly effective method of contraception, if of childbearing potential and has a negative urine human chorionic gonadotropin beta subunit (B-HCG) pregnancy test during screening, and prior to trial drug administration.

Exclusion Criteria:

1. Subjects already on or failed omeprazole in past, or intolerant of PPI therapy
2. Subjects who are using clopidogrel (Plavix)
3. Subjects with one or more of the following diagnoses:

   1. Neoplasm of the esophagus or stomach
   2. Previous upper gastrointestinal surgery (esophagectomy, Heller myotomy, hiatal hernial repair)
   3. Diabetic gastroparesis
   4. Esophageal motility disorder: Achalasia or scleroderma
   5. Zollinger-Ellison syndrome
   6. Infection with human immunodeficiency virus (HIV)
   7. Bleeding diathesis
   8. History of gastric or small bowel obstruction
   9. Inability to read due to blindness, cognitive dysfunction, English language illiteracy
   10. Disorders which predispose to unreliable responses such as Schizophrenia, Alzheimer's disease or significant memory loss
   11. Pregnant and lactating females will be excluded as PPIs are not thought safe for the fetus (Pregnancy Category C).
4. Children younger than 18 years of age will be excluded as their compliance might be dictated by others, such as their parents, and their results would not be generalizable to the adult population. Other vulnerable populations, such as those with diminished mental acuity, will be excluded for the same reason.
5. Residence outside of the US (due to difficulties with overseas postal service) or in prison.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Romero, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Mayo Clinic in Rochester, MN from June 20, 2008 to May 24, 2010.
Pre-assignment Details: One subject on the PM dose arm did not receive allocated intervention because the subject changed their mind soon after randomization.
Period: Overall Study
Arm/Group | Omeprazole/Sodium Bicarbonate AM Dose | Omeprazole/Sodium Bicarbonate PM Dose
Started | 43 | 48
Completed | 41 | 43
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 1 | 2
Not completed — Adverse Event | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omeprazole/Sodium Bicarbonate AM Dose | Omeprazole/Sodium Bicarbonate PM Dose | Total
Number analyzed (Participants) | 43 | 48 | 91
Age Continuous [Mean (Full Range); unit: years] | 58 [19 to 86] | 59 [30 to 86] | 58 [19 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 30 | 33 | 63
Region of Enrollment [Number; unit: participants]
  United States | 43 | 48 | 91
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 31.1 [24.5 to 51] | 31.1 [21.2 to 46.8] | 31.1 [21.2 to 51]
Esophagitis Severity [Number; unit: participants] — Esophagitis Severity was measured in Los Angeles (LA) Classification system, which quantifies erosive esophagitis and is graded on an A-D scale with increasing severity of injury.
  participants
    LA grade C (moderate esophagitis) | 26 | 33 | 59
    LA grade D (severe esophagitis) | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Overall Who Healed, Improved, or Stayed the Same or Worsened After 8 Weeks of Treatment
Description: After 8 weeks of treatment a follow-up esophagogastroduodenoscopy (EGD) was performed by an endoscopist blinded to the study and subject allocation. The evaluation results were grouped as follows:
  LA C esophagitis at baseline: healed = no erosions in the esophagus; improved= LA grades A or B; Same or worse = C or D at follow-up LA D esophagitis at baseline: healed = no erosions in the esophagus; improved=LA grades A, B, or C; Same=LA grade D at follow-up.
Time Frame: 8 weeks
Measure: Number; unit: percentage of patients
Arm/Group | Omeprazole/Sodium Bicarbonate AM Dose | Omeprazole/Sodium Bicarbonate PM Dose
Number analyzed (Participants) | 41 | 43
percentage of patients
  Healed | 83 | 81
  Improved | 15 | 14
  Same or worse | 2 | 5
Statistical Analysis 1: Comparison: Omeprazole/Sodium Bicarbonate AM Dose vs Omeprazole/Sodium Bicarbonate PM Dose; Test type: Superiority or Other; p = 1.0, Fisher Exact

2. Secondary Outcome: Percent of Subjects With Moderate Esophagitis (LA Grade C) Who Healed, Improved, or Stayed the Same or Worsened After 8 Weeks of Treatment
Description: as for outcome 1
Time Frame: 8 weeks
Population: 25 of the 41 participants in the Omeprazole/sodium bicarbonate AM dose arm were LA Grade C. 29 of the 43 participants in the Omeprazole/sodium bicarbonate AM dose arm were LA Grade C.
Measure: Number; unit: percentage of participants
Arm/Group | Omeprazole/Sodium Bicarbonate AM Dose | Omeprazole/Sodium Bicarbonate PM Dose
Number analyzed (Participants) | 25 | 29
percentage of participants
  Healed | 88 | 79
  Improved | 12 | 14
  Same or worse | 0 | 7

3. Secondary Outcome: Percent of Subjects With Severe Esophagitis (LA Grade D) Who Healed, Improved, or Stayed the Same After 8 Weeks of Treatment
Description: as for outcome 1
Time Frame: 8 weeks
Population: 16 of the 41 participants in the Omeprazole/sodium bicarbonate AM dose arm were LA Grade D. 14 of the 43 participants in the Omeprazole/sodium bicarbonate PM dose arm were LA Grade D.
Measure: Number; unit: percentage of participants
Arm/Group | Omeprazole/Sodium Bicarbonate AM Dose | Omeprazole/Sodium Bicarbonate PM Dose
Number analyzed (Participants) | 16 | 14
percentage of participants
  Healed | 75 | 86
  Improved | 19 | 14
  Same | 6 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the eight weeks subjects were on study drug.
Arm/Group | Omeprazole/Sodium Bicarbonate AM Dose | Omeprazole/Sodium Bicarbonate PM Dose
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/43
Other Adverse Events (participants affected / at risk) | 1/41 | 3/43
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omeprazole/Sodium Bicarbonate AM Dose (N=41) | Omeprazole/Sodium Bicarbonate PM Dose (N=43)
Joint and muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
peripheral edema/increased blood pressue (Blood and lymphatic system disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Our methods relied upon pill counting as a proxy for adherence to medical therapy. Now that PPIs are available over the counter, few patients present de novo with LA C and LA D esophagitis. We didn't control for other factors that can affect GERD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No